CLINICAL TRIAL: NCT03527836
Title: Comparison of Plasma Concentrations of Lidocaine and Bupivacaine After Ultrasound-guided Axillary Approach to Brachial Plexus Block Used With Different Dilute Mixture Solutions for Upper Limb Trauma Surgery
Brief Title: Plasma Concentration of Lidocaine and Bupivacaine Axillary BPB Mixture Solutions [PCLBAxMix]
Acronym: PCLBAxMix
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 6634
Record Dates: First submitted 2018-02-15; First posted 2018-05-17 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Arm Injury
MeSH Terms: conditions — Arm Injuries | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Study participants n=10 in the L group, n=10 in the B group and n=10 in the mixture group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients, the operating team, nurses, and observers involved in the assessment of the follow-up data collection were unaware of group allocation. The labor analyst is unaware of group allocation.
  The list of cases will be provided in spreadsheet program by an observer-blinded assistant and was statistically evaluated by an independent analyst.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lidocaine (Active Comparator): Lidocaine brachial plexus block 0.4 ml/kg of 0.66% solution
  Interventions: Drug: Lidocaine brachial plexus block
- Bupivacaine (Active Comparator): Bupivacaine brachial plexus block 0.4 ml/kg of 0.33% solution
  Interventions: Drug: Bupivacaine brachial plexus block
- Mixture (Active Comparator): Mixture brachial plexus block 0.4 ml/kg of 0.33% bupivacaine and 0.33% lidocaine solution
  Interventions: Drug: Mixture brachial plexus block

INTERVENTIONS:
Drug: Lidocaine brachial plexus block — Combined Axillary-supraclavicular approach to brachial plexus with lidocaine
  Other Names: Lidocain-EGIS 1% OGYI-T-3047/03
  Arms: Lidocaine
Drug: Bupivacaine brachial plexus block — Combined Axillary-supraclavicular approach to brachial plexus with bupivacaine
  Other Names: Marcaine 5 mg/ml Astra Zeneca OGYI-T 6496/14
  Arms: Bupivacaine
Drug: Mixture brachial plexus block — Combined Axillary-supraclavicular approach to brachial plexus with mixture solution of 20 ml bupivacaine 0.5% and 10 ml lidocaine 1%
  Other Names: Lidocain-EGIS 1% and Marcaine 5 mg/ml Astra Zeneca
  Arms: Mixture

SUMMARY:
The doses of local anesthetics can be decreased with the use of ultrasound guidance. In case of using mixture solutions the benefits and drawbacks are controversial. The plasma concentrations were not studied up to this time in this kind of settings, so investigators believe that this is the first work that shows how lidocaine change the plasma concentration of bupivacaine after axillary approach to brachial plexus employed with different dilute and mixed solutions for upper limb surgery in trauma patients.

DETAILED DESCRIPTION:
Total of 30 American Society of Anesthesiologist (ASA) I-III adult patients scheduled to elective or emergency trauma surgery of hand and forearm under ultrasound-guided (UG) brachial plexus block (BPB) are planned to be assigned into this randomized-prospective observational study after approval by the University Research Ethics Board, Pécs University Medical School, Hungary. All of the patients will receive detailed information about the planned BPB techniques and surgeries, then written informed consents will be obtained.

Study participants are planned to be assigned randomly by the research coordinator into 3 groups (Lidocaine, Bupivacaine and mixture solution) according to the concentration of lidocaine and bupivacaine in the mixture solution.

Standardized UG Axillary-supraclavicular (AX-SC) approach to the BP is planned to be performed under sterile conditions by the same anesthesiologist. The standardized dose is 0.4 ml/kg with the targeted maximized the single-shot volume of 30 ml.

Blood samples will be taken at 0-time point (straight after the administration of BP injection) and 30, 60, 240 and 480 minutes after. Plasma concentrations are determined, the results are collected and analyzed.

Under standard monitorization, vital parameters, data are collected on the onset time and duration of actions of local anesthetics (LAs).

ELIGIBILITY:
Inclusion Criteria:

* unpremedicated patient scheduled for elective or emergency trauma surgery of hand and forearm under ultrasound-guided BPB

Exclusion Criteria:

* continuous peripheral nerve catheter technique or bilateral block was planned, or the patient refused to participate. Exclusion criteria included psycho-mental conditions interfering with consent or assessment; pre-existing chronic pain condition or daily analgesic or sedative consumption; sedative or analgesic premedication; pre-existing neurological disorders aﬀecting the brachial plexus.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-17 (Actual); Primary Completion 2021-12-17 (Estimated); Study Completion 2022-01-17 (Estimated)

PRIMARY OUTCOMES:
Maximal plasma concentrations | 0-8 hours
  Plasma concentrations of bupivacaine and lidocaine 0-8 hours after injection

SECONDARY OUTCOMES:
Onset times | 0-0.5 hours
  Onset times of local anesthetics
Duration | 1-24 hours
  Duration of actions of local anesthetics

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Almasi, PhD. habil, Study Chair — University of Pecs, Medical School, Pain Medicine Dept.of Anesth Int Care; Barbara Rezman, MD, Principal Investigator — University of Pecs, Medical School, Dept.of Anesth Int Care
Locations (1):
- University of Pécs, Medical School, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: No